CLINICAL TRIAL: NCT00875823
Title: International Registry for Hereditary Calcium Stone Diseases
Brief Title: International Registry for Primary Hyperoxaluria
Status: Withdrawn | Type: Observational
Why Stopped: Study was combined with Mayo protocol 07-003476
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Oxalosis and Hyperoxaluria Foundation (OHF) (Other)
Responsible Party: John C. Lieske, M.D., Mayo Clinic Department of Nephrology
Other Study IDs: 1605-03; NCT00616525 (obsolete NCT alias)
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Primary Hyperoxaluria; Nephrocalcinosis; Kidney Stones
Keywords: PH; Primary Hyperoxaluria; Type I; Type II; NonI-NonII; Kidney stones; oxalate; oxalosis
MeSH Terms: conditions — Hyperoxaluria, Primary; Nephrocalcinosis; Kidney Calculi; Hyperoxaluria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PH Patients: Patients with:
  Primary Hyperoxaluria Type I Primary Hyperoxaluria Type II Primary Hyperoxaluria NonI-NonII

SUMMARY:
The purpose of this study is to collect medical information from a large number of patients in many areas of the world with primary hyperoxaluria. This medical information will be entered into a registry to help the investigators compare similarities and differences in patients and their symptoms. The more patients that the investigators are able to enter into the registry, the more the investigators will be able to understand primary hyperoxaluria and learn better ways of treating patients with this disease. It is the investigators hope that by entering as many patients with PH as possible, the information that the investigators collect may help physicians diagnose patients sooner and determine what treatments may work best on patients with similar medical or genetic backgrounds.

DETAILED DESCRIPTION:
This study involves the collection of medical information to create a computer database (registry) for patients with PH. The information will be entered into the registry by your physician, healthcare provider or a staff member of the Mayo Clinic Hyperoxaluria Center. The computer web site for the registry is secure and protected by a required password. Some information which will be entered may include your age at first symptoms of PH,kidney stone history, lab values, kidney function, and your health over time. Information for a patient can only be viewed by the appropriate physician and staff. Once the information is entered into the registry, you will only be identified by a code number.

ELIGIBILITY:
Inclusion Criteria:

* Liver biopsy or genetic analysis that confirms a diagnosis of hyperoxaluria
* In the absence of a liver biopsy:
* Urine oxalate excretion of >0.8 mmol/1.73 m² /day without other causes such as enteric hyperoxaluria
* Family history of PH in a sibling will be supportive
* A history or current finding of kidney stones or nephrocalcinosis will be supportive
* An increase in urine glycolate may suggest PHI or an increase in urine L-glycerate may suggest PHII, though not required for diagnosis.
* Patients presenting in renal failure with an elevate pre-dialysis plasma oxalate of 60 umol/l and a kidney biopsy that confirms extensive oxalate deposition, or evidence of systemic oxalosis

Exclusion Criteria:

* Patients without any of the above or a confirmed diagnosis of PH

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with a confirmed diagnosis of primary hyperoxaluria (PH)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2003-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Lieske, M.D., Principal Investigator — Mayo Clinic Department of Nephrology and Hypertension
Locations (4):
- United States (4):
  - Mattel Children's Hospital at UCLA, Los Angeles, California
  - University of California at Davis, Sacramento, California
  - Children's Memorial Hospital, Chicago, Illinois
  - Mayo Clinic Rochester, Rochester, Minnesota

REFERENCES:
- [Result] Lieske JC, Monico CG, Holmes WS, Bergstralh EJ, Slezak JM, Rohlinger AL, Olson JB, Milliner DS. International registry for primary hyperoxaluria. Am J Nephrol. 2005 May-Jun;25(3):290-6. doi: 10.1159/000086360. Epub 2005 Jun 15. PMID 15961949
- See also: Mayo Clinic Hyperoxaluria Center — http://www.mayoclinic.org/nephrology-rst/hyperoxaluriacenter.html
- See also: Oxalosis and Hyperoxaluria Foundation — http://www.ohf.org